CLINICAL TRIAL: NCT00759564
Title: An Open-label, 2-way Crossover Study To Investigate The Pharmacokinetics, Safety And Tolerability Of Iv Cp-70429 And Oral Pf-03709270 In Subjects With Varying Degrees Of Renal Impairment And Normal Renal Function
Brief Title: A Study To Investigate The Pharmacokinetics, Safety And Tolerability Of An Intravenous And Oral Form Of A Compound In Subjects With Varying Degrees Of Renal Impairment And Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: A8811009; 2009-017796-20 (EudraCT Number)
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — sulopenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV CP-70,429 and cross over to PF-03709270 (Experimental)
  Interventions: Drug: CP-70,429 and PF-03709270

INTERVENTIONS:
Drug: CP-70,429 and PF-03709270 — Study Periods 1 and 2 will be separated by a minimum of 14 days. In Period 1, subjects will receive a single dose of CP-70429 (800 mg given as a 1.5 hour intravenous infusion), while in Period 2, subjects will receive a single oral dose of PF-03709270 (1000 mg).
  Other Names: CP-70,429 - sulopenem

SUMMARY:
This study will evaluate what effect renal dysfunction has on a drug that has an intravenous (CP-70,429) and an oral form (PF-03709270).

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics and safety.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet one of the following renal function categories:

* Normal renal function (CLcr >80 mL/min).
* Mild renal impairment (CLcr >50 and <80 mL/min).
* Moderate renal impairment (CLcr >30 and <50 mL/min).
* Severe renal impairment (CLcr <30 mL/min).

Exclusion Criteria:

Women who are pregnant or nursing or women who are of childbearing potential. History of clinically significant allergies, including seasonal allergies, and especially drug hypersensitivity including known allergies to components of the study drug formulation, penicillin, carbapenems and/or cephalosporin antibiotics (eg, amoxicillin, amoxicillin/clavulanate, ampicillin, cefadroxil, cephalexin, cefaclor and cefixime).

Subjects should not have evidence of a history of the following:

* normal renal function: clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological or allergic disease.
* renal impairment: any clinically significant (hepatic, cardiac or pulmonary or subjects with acute nephritic syndrome) diseases (except diabetes). Stable co-morbid disease where it is unlikely that the disease and medication will alter the outcome of the study will be allowed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Centurion Clinical Research, Indianapolis, Indiana, United States
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8811009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a fixed sequence design study (not a complete 2 way crossover) in parallel groups of participants with varying degrees of renal impairment, where all subjects received the intravenous formulation in first period and then received the oral formulation in second period.
Pre-assignment Details: Participants were planned to receive CP-70,429 800 milligram (mg) in all reporting groups. For severe renal impairment group, CP-70,429 dose was decreased from 800 mg to 200 mg as per protocol amendment. Only 1 participant received 800 mg dose and was excluded from all descriptive and statistical analyses as per change in planned analysis.
Groups:
- CP-70,429 (800 mg) + PF-03709270: Normal Renal Function: Participants with normal renal function (defined by creatinine clearance [CLcr] greater than [>] 80 milliliter per minute [mL/min]) received a single dose of CP-70,429 800 mg given as an intravenous infusion over 1.5 hours in first intervention period followed by a single oral dose of PF-03709270 1000 mg in second intervention period. A washout period of at least 14 days was maintained between each intervention period.
- CP-70,429 (800 mg) + PF-03709270: Mild Renal Impairment: Participants with mild renal impairment (defined by CLcr >50 and less than or equal to [<=] 80 mL/min) received a single dose of CP-70,429 800 mg given as an intravenous infusion over 1.5 hours in first intervention period followed by a single oral dose of PF-03709270 1000 mg in second intervention period. A washout period of at least 14 days was maintained between each intervention period.
- CP-70,429 (800 mg) + PF-03709270: Moderate Renal Impairment: Participants with moderate renal impairment (defined by CLcr greater than or equal to >=30 and <=50 mL/min) received a single dose of CP--70,429 800 mg given as an intravenous infusion over 1.5 hours in first intervention period followed by a single oral dose of PF-03709270 1000 mg in second intervention period. A washout period of at least 14 days was maintained between each intervention period.
- CP-70,429 (800 mg) + PF-03709270: Severe Renal Impairment: Participants with severe renal impairment (defined by CLcr <30 mL/min) received a single dose of CP-70,429 800 mg given as an intravenous infusion over 1.5 hours in first intervention period followed by a single oral dose of PF-03709270 1000 mg in second intervention period. A washout period of at least 14 days was maintained between each intervention period.
- CP-70,429 (200 mg) + PF-03709270: Severe Renal Impairment: Participants with severe renal impairment (defined by CLcr <30 mL/min) received a single dose of CP--70,429 200 mg given as an intravenous infusion over 1.5 hours in first intervention period followed by a single oral dose of PF--03709270 1000 mg in second intervention period. A washout period of at least 14 days was maintained between each intervention period.
Period: First Intervention Period (4 Days)
Arm/Group | CP-70,429 (800 mg) + PF-03709270: Normal Renal Function | CP-70,429 (800 mg) + PF-03709270: Mild Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Moderate Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Severe Renal Impairment | CP-70,429 (200 mg) + PF-03709270: Severe Renal Impairment
Started | 8 | 8 | 8 | 1 | 4
Completed | 8 | 8 | 8 | 1 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | CP-70,429 (800 mg) + PF-03709270: Normal Renal Function | CP-70,429 (800 mg) + PF-03709270: Mild Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Moderate Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Severe Renal Impairment | CP-70,429 (200 mg) + PF-03709270: Severe Renal Impairment
Started | 8 | 8 | 8 | 1 | 4
Completed | 8 | 8 | 8 | 1 | 3
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Second Intervention Period (4 Days)
Arm/Group | CP-70,429 (800 mg) + PF-03709270: Normal Renal Function | CP-70,429 (800 mg) + PF-03709270: Mild Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Moderate Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Severe Renal Impairment | CP-70,429 (200 mg) + PF-03709270: Severe Renal Impairment
Started | 8 | 8 | 8 | 1 | 3
Completed | 8 | 8 | 8 | 1 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CP-70,429 (800 mg) + PF-03709270: Normal Renal Impairment: Participants with normal renal function (defined by creatinine clearance [CLcr] greater than [>] 80 milliliter per minute [mL/min]) received a single dose of CP-70,429 200 mg given as an intravenous infusion over 1.5 hours in first intervention period followed by a single oral dose of PF-03709270 1000 mg in second intervention period. A washout period of at least 14 days was maintained between each intervention period.
- CP-70,429 (200 mg) + PF-03709270: Severe Renal Function: Participants with severe renal impairment (defined by CLcr <30 mL/min) received a single dose of CP--70,429 200 mg given as an intravenous infusion over 1.5 hours in first intervention period followed by a single oral dose of PF--03709270 1000 mg in second intervention period. A washout period of at least 14 days was maintained between each intervention period.
- Total: Total of all reporting groups
Arm/Group | CP-70,429 (800 mg) + PF-03709270: Normal Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Mild Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Moderate Renal Impairment | CP-70,429 (800 mg) + PF-03709270: Severe Renal Impairment | CP-70,429 (200 mg) + PF-03709270: Severe Renal Function | Total
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 4 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (3.2) | 60.6 (7.3) | 64.3 (15.7) | 55 (NA) — Standard deviation was not calculated as single participant was analyzed. | 69 (9.4) | 62.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 0 | 4 | 12
  Male | 5 | 5 | 6 | 1 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of CP-70429 Following CP-70,429 Intravenous Dose
Description: PF-03709270 is an oral prodrug of CP-70,429. Upon oral absorption, PF-03709270 is rapidly hydrolyzed, yielding the active drug CP-70,429. Cmax of CP-70429 following CP-70,429 intravenous dose was reported.
Time Frame: 0 (pre-dose), 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose (for all participants) and 48 hours post-dose (for participants with moderate and severe renal impairment)
Population: The pharmacokinetic (PK) parameter analysis population included all treated participants who had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- CP-70,429 (800 mg): Normal Renal Function: Participants with normal renal function (defined by CLcr >80 mL/min) received a single dose of CP-70,429 800 mg given as an intravenous infusion over 1.5 hours in first intervention period.
- CP-70,429 (800 mg): Mild Renal Impairment: Participants with mild renal impairment (defined by CLcr >50 and <=80 mL/min) received a single dose of CP-70,429 800 mg given as an intravenous infusion over 1.5 hours in first intervention period.
- CP-70,429 (800 mg): Moderate Renal Impairment: Participants with moderate renal impairment (defined by CLcr >=30 and <=50 mL/min) received a single dose of CP-70,429 800 mg given as an intravenous infusion over 1.5 hours in first intervention period.
- CP-70,429 (200 mg): Severe Renal Impairment: Participants with severe renal impairment (defined by CLcr <30 mL/min) received a single dose of CP-70,429 200 mg given as an intravenous infusion over 1.5 hours in first intervention period.
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
nanogram per milliliter (ng/mL) | 17700 (1880.3) | 22070 (3420.8) | 28940 (6880.0) | 10340 (2784.3)
Statistical Analysis 1: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (800 mg): Mild Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed Cmax for mild renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 124.71, 90% CI 2-sided [106.57 to 145.94]
Statistical Analysis 2: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (800 mg): Moderate Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed Cmax for moderate renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 163.51, 90% CI 2-sided [139.72 to 191.34]
Statistical Analysis 3: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (200 mg): Severe Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed Cmax for severe renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 58.40, 90% CI 2-sided [48.16 to 70.83]

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of CP-70429 Following CP-70,429 Intravenous Dose
Time Frame: as for outcome 1
Population: The PK parameter analysis population included all treated participants who had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Median (Full Range); unit: hours
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 1.00 (11) [1.00 to 1.50] | 1.50 (15) [1.00 to 1.50] | 1.50 (23) [1.50 to 1.50] | 1.50 (26) [1.00 to 1.50]

3. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of CP-70429 Following CP-70,429 Intravenous Dose
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the time of last measured concentration (AUClast).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
nanogram*hour per milliliter (ng*hr/mL) | 31990 (4793.3) | 53610 (10520) | 78940 (23937) | 34270 (8430.3)
Statistical Analysis 1: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (800 mg): Mild Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed AUClast for mild renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 167.59, 90% CI 2-sided [137.27 to 204.61]
Statistical Analysis 2: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (800 mg): Moderate Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed AUClast for moderate renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 246.76, 90% CI 2-sided [202.11 to 301.27]
Statistical Analysis 3: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (200 mg): Severe Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed AUClast for severe renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 107.13, 90% CI 2-sided [88.06 to 130.32]

4. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-inf)] of CP-70,429 Following CP-70,429 Intravenous Dose
Description: AUC (0-inf) is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng*hr/mL | 32160 (4775.5) | 54070 (10647) | 79870 (24619) | 35410 (9610.6)
Statistical Analysis 1: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (800 mg): Mild Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed AUCinf for mild renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 168.14, 90% CI 2-sided [137.40 to 205.75]
Statistical Analysis 2: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (800 mg): Moderate Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed AUCinf for moderate renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 248.38, 90% CI 2-sided [202.98 to 303.94]
Statistical Analysis 3: Comparison: CP-70,429 (800 mg): Normal Renal Function vs CP-70,429 (200 mg): Severe Renal Impairment; A one-way ANOVA model with group as a fixed effect was used to compare the natural log transformed AUCinf for severe renal impairment group (Test) to normal renal function group (Reference). The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Percent Geometric Mean Ratio = 110.12, 90% CI 2-sided [89.84 to 134.98]

5. Primary Outcome: Renal Clearance (CLr) of CP-70429 Following CP-70,429 Intravenous Dose
Description: Renal clearance was calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Ae) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau).
Time Frame: 0 (pre-dose), 0 to 6, 6 to 12, 12 to 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
liter per hour (L/hr) | 8.035 (5.578) | 6.936 (2.516) | 3.043 (3.297) | 2.303 (0.605)

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of CP-70429 Following PF-03709270 Oral Dose
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- PF--03709270 (1000 mg): Normal Renal Function: Participants with normal renal function (defined by CLcr >80 mL/min) received a single oral dose of PF--03709270 1000 mg tablet in second intervention period.
- PF--03709270 (1000 mg): Mild Renal Impairment: Participants with mild renal impairment (defined by CLcr >50 and <=80 mL/min) received a single oral dose of PF--03709270 1000 mg tablet in second intervention period.
- PF--03709270 (1000 mg): Moderate Renal Impairment: Participants with moderate renal impairment (defined by CLcr >=30 and <=50 mL/min) received a single oral dose of PF--03709270 1000 mg tablet in second intervention period.
- PF--03709270 (1000 mg): Severe Renal Impairment: Participants with severe renal impairment (defined by CLcr <30 mL/min) received a single oral dose of PF--03709270 1000 mg tablet in second intervention period.
Arm/Group | PF--03709270 (1000 mg): Normal Renal Function | PF--03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF--03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng/mL | 2747 (420.58) | 3704 (1053.3) | 6215 (1841.3) | 7830 (738.17)
Statistical Analysis 1: Comparison: PF--03709270 (1000 mg): Normal Renal Function vs PF--03709270 (1000 mg): Mild Renal Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 134.86, 90% CI 2-sided [109.88 to 165.52]
Statistical Analysis 2: Comparison: PF--03709270 (1000 mg): Normal Renal Function vs PF--03709270 (1000 mg): Moderate Renal Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 226.28, 90% CI 2-sided [184.36 to 277.72]
Statistical Analysis 3: Comparison: PF--03709270 (1000 mg): Normal Renal Function vs PF--03709270 (1000 mg): Severe Renal Impairment; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 285.05, 90% CI 2-sided [221.80 to 366.33]

7. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of CP-70429 Following PF-03709270 Oral Dose
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Groups:
- PF--03709270 (1000 mg): Mild Renal Impairment: Participants with mild renal impairment (defined by CLcr >50 and <=80 mL/min) received a single oral dose of PF-03709270 1000 mg tablet in second intervention period.
Arm/Group | PF--03709270 (1000 mg): Normal Renal Function | PF--03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF--03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 1.50 (11) [0.50 to 2.00] | 2.50 (15) [1.00 to 4.00] | 1.50 (23) [1.00 to 3.00] | 2.50 (26) [1.50 to 4.00]

8. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of CP-70429 Following PF-03709270 Oral Dose
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- PF-03709270 (1000 mg): Normal Renal Function: Participants with normal renal function (defined by CLcr >80 mL/min) received a single oral dose of PF--03709270 1000 mg tablet in second intervention period.
- PF-03709270 (1000 mg): Severe Renal Impairment: Participants with severe renal impairment (defined by CLcr <30 mL/min) received a single oral dose of PF-03709270 1000 mg tablet in second intervention period.
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF--03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng*hr/mL | 6403 (1355.9) | 13400 (4948.8) | 22600 (9034.3) | 47560 (15782)
Statistical Analysis 1: Comparison: PF-03709270 (1000 mg): Normal Renal Function vs PF--03709270 (1000 mg): Mild Renal Impairment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 209.31, 90% CI 2-sided [158.81 to 275.87]
Statistical Analysis 2: Comparison: PF-03709270 (1000 mg): Normal Renal Function vs PF--03709270 (1000 mg): Moderate Renal Impairment; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 353.00, 90% CI 2-sided [267.83 to 465.25]
Statistical Analysis 3: Comparison: PF-03709270 (1000 mg): Normal Renal Function vs PF-03709270 (1000 mg): Severe Renal Impairment; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 742.68, 90% CI 2-sided [529.59 to 1041.50]

9. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-inf)] of CP-70429 Following PF-03709270 Oral Dose
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF--03709270 (1000 mg): Normal Renal Function | PF--03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
ng*hr/mL | 6523 (1329.5) | 13670 (5088.1) | 23040 (9403.9) | 47990 (16191)
Statistical Analysis 1: Comparison: PF--03709270 (1000 mg): Normal Renal Function vs PF--03709270 (1000 mg): Mild Renal Impairment; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 209.55, 90% CI 2-sided [158.72 to 276.66]
Statistical Analysis 2: Comparison: PF--03709270 (1000 mg): Normal Renal Function vs PF--03709270 (1000 mg): Moderate Renal Impairment; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 353.26, 90% CI 2-sided [267.57 to 466.39]
Statistical Analysis 3: Comparison: PF--03709270 (1000 mg): Normal Renal Function vs PF-03709270 (1000 mg): Severe Renal Impairment; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; Percent Geometric Mean Ratio = 735.77, 90% CI 2-sided [523.56 to 1034.00]

10. Primary Outcome: Renal Clearance (CLr) of CP-70429 Following PF-03709270 Oral Dose
Description: as for outcome 5
Time Frame: 0 (pre-dose), 0 to 6, 6 to 12, 12 to 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Groups:
- PF-03709270 (1000 mg): Normal Renal Function: Participants with normal renal function (defined by CLcr >80 mL/min) received a single oral dose of PF-03709270 1000 mg tablet in second intervention period.
- PF-03709270 (1000 mg): Mild Renal Impairment: Participants with mild renal impairment (defined by CLcr >50 and <=80 mL/min) received a single oral dose of PF-03709270 1000 mg tablet in second intervention period.
- PF--03709270: Severe Renal Impairment: Participants with severe renal impairment (defined by CLcr <30 mL/min) received a single oral dose of PF--03709270 1000 mg tablet in second intervention period.
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF--03709270: Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
L/hr | 15.47 (1.885) | 7.952 (2.537) | 4.239 (2.647) | 3.294 (4.398)

11. Secondary Outcome: Terminal Elimination Half Life (t1/2) of CP-70429 Following CP-70,429 Intravenous Dose
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 1.034 (0.216) | 1.660 (0.586) | 1.823 (0.269) | 2.313 (0.579)

12. Secondary Outcome: Terminal Elimination Half Life (t1/2) of CP-70429 Following PF-03709270 Oral Dose
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF--03709270: Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 0.837 (0.121) | 1.451 (0.335) | 1.809 (0.566) | 2.750 (0.832)

13. Secondary Outcome: Clearance (CL)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. It was calculated by dividing given intravenous dose by AUC inf. AUC inf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
L/hr | 24.87 (3.9001) | 14.79 (2.6787) | 10.01 (3.7432) | 5.648 (1.2500)

14. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. It was calculated by dividing the given oral dose by AUCinf. AUC inf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Groups:
- PF-03709270 (1000 mg): Moderate Renal Impairment: Participants with moderate renal impairment (defined by CLcr >=30 and <=50 mL/min) received a single oral dose of PF-03709270 1000 mg tablet in second intervention period.
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
L/hr | 153.5 (31.540) | 73.20 (24.115) | 43.38 (19.719) | 20.86 (6.8699)

15. Secondary Outcome: Duration of Plasma Concentrations of CP-70429 Exceeding 0.5 Microgram Per Milliliter Following Intravenous Dose
Description: Duration was calculated by subtracting the time at which the plasma concentrations exceeded 0.5 microgram per milliliter (mcg/mL) at the ascending part of the concentration-time profile from the time at which the plasma concentrations fell below 0.5 mcg/mL at the descending part of the profile. If these times fell between 2 observed concentrations, a method of linear interpolation was used for best estimation.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 5.310 (0.641) [3.93 to 5.56] | 8.855 (1.542) [6.23 to 11.1] | 11.40 (3.389) [6.67 to 16.8] | 10.70 (4.009) [6.65 to 16.4]

16. Secondary Outcome: Duration of Plasma Concentrations of CP-70429 Exceeding 0.5 Microgram Per Milliliter Following PF-03709270 Oral Dose
Description: Duration was calculated by subtracting the time at which the plasma concentrations exceeded 0.5 mcg/mL at the ascending part of the concentration-time profile from the time at which the plasma concentrations fell below 0.5 mcg/mL at the descending part of the profile. If these times fell between 2 observed concentrations, a method of linear interpolation was used for best estimation.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF--03709270: Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 3.915 (0.121) [2.76 to 4.88] | 6.440 (0.335) [5.03 to 10.9] | 8.185 (0.566) [5.60 to 11.7] | 18.30 (0.832) [9.48 to 22.0]

17. Secondary Outcome: Duration of Plasma Concentrations of CP-70429 Exceeding 1.0 Microgram Per Milliliter Following Intravenous Dose
Description: Duration was calculated by subtracting the time at which the plasma concentrations exceeded 1.0 mcg/mL at the ascending part of the concentration-time profile from the time at which the plasma concentrations fell below 1.0 mcg/mL at the descending part of the profile. If these times fell between 2 observed concentrations, a method of linear interpolation was used for best estimation.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 3.935 (0.461) [3.32 to 4.69] | 7.190 (0.849) [5.50 to 7.88] | 9.240 (2.161) [5.65 to 11.6] | 7.710 (2.304) [5.52 to 11.1]

18. Secondary Outcome: Duration of Plasma Concentrations of CP-70429 Exceeding 1.0 Microgram Per Milliliter Following PF-03709270 Oral Dose
Description: as for outcome 16
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF--03709270 (1000 mg): Moderate Renal Impairment | PF--03709270: Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours | 2.895 (0.121) [1.95 to 3.42] | 4.990 (0.335) [3.29 to 8.66] | 6.320 (0.566) [4.47 to 9.72] | 12.15 (0.832) [7.38 to 19.4]

19. Secondary Outcome: Pharmacokinetics of CP-70429 and PF-03709270 Metabolites
Description: PF-03709270 is an oral prodrug of CP-70,429. Upon oral absorption, PF-03709270 is rapidly hydrolyzed, yielding the active drug CP-70,429 and metabolites.
Time Frame: 0.5, 2, 4, 8, 12, 24 hours post-dose (for all participants) and 48 hours post-dose (for participants with moderate and severe renal impairment)
Population: Data was not collected for this outcome because the metabolite data for CP-70,429 and PF-03709270 were not analyzed as per change in planned analysis
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Concentration Versus Time Summary of 2-Ethylbutyric Acid
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLQ =100 ng/mL) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) =0.
Time Frame: 1, 3, 8 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours
  1 hour | 46.38 (96.048) | 19.00 (53.740) | 15.25 (43.134) | NA (NA) — No observations above the lower limit of quantification.
  3 hours | 20.00 (56.569) | 17.63 (49.851) | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification.
  8 hours | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification.

21. Secondary Outcome: Concentration Versus Time Summary of Plasma Formate
Description: as for outcome 20
Time Frame: 1, 3, 8 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 4
hours
  1 hour | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification.
  3 hours | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification.
  8 hours | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification. | NA (NA) — No observations above the lower limit of quantification.

22. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 7-10 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 7-10 days after the last dose of study drug (up to 32 days)
Population: Safety analysis set included all participants who received the study medication.
Measure: Number; unit: participants
Groups:
- CP-70,429 (800 mg): Severe Renal Impairment: Participants with severe renal impairment received a single dose of CP-70,429 800 mg given as a 1.5-hour intravenous infusion under fasted condition in first intervention period.
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (800 mg): Severe Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 4 | 8 | 8 | 8 | 4
participants
  AEs | 5 (0.216) | 5 (0.586) | 4 (0.269) | 0 (0.579) | 3 (0.121) | 6 (0.335) | 4 (0.566) | 6 (0.831) | 3
  SAEs | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory test abnormality: Hematology (hemoglobin, hematocrit, red blood corpuscles [RBC] count: less than [<]0.8*lower limit of normal [LLN], platelets: <0.5*LLN/greater than [>]1.75*upper limit of normal [ULN], leukocytes: <0.6*LLN or >1.5*ULN, lymphocytes, total neutrophils: <0.8*LLN or >1.2*ULN, basophils, eosinophil, monocytes: >1.2*ULN); Liver Function (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >0.3*ULN, total protein, albumin: <0.8*LLN or >1.2*ULN); total bilirubin, direct bilirubin, indirect bilirubin: >1.5*ULN; Renal Function (blood urea nitrogen, creatinine: >1.3*ULN, uric acid: >1.2*ULN); Electrolytes (sodium: <0.95*LLN or >1.05*ULN, potassium, chloride, calcium, bicarbonate: <0.9*LLN or >1.1*ULN; creatine kinase: >2.0*ULN; glucose fasting: <0.6*LLN or >1.5*ULN, urine white blood corpuscles [WBC] and RBC: greater than or equal to (>=) 6/High Power Field [HPF]).
Time Frame: Baseline up to 7-10 days after the last dose of study drug (up to 32 days)
Population: Safety analysis set included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (800 mg): Severe Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 4 | 8 | 8 | 8 | 4
participants | 2 | 3 | 7 | 1 | 4 | 1 | 3 | 8 | 4

24. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Criteria for vital signs abnormalities included supine/sitting pulse rate of <40 beats per minute (bpm) or >120 bpm, supine systolic blood pressure (SBP) of <90 millimeter of mercury (mmHg), >=30 mmHg maximum increase and decrease from baseline in same posture, supine diastolic blood pressure (DBP) of <50 mmHg, >=20 mmHg maximum increase and decrease from baseline in same posture, heart rate <=45 beats per minute (bpm) or >=120 bpm or decrease/increase of >=15 bpm.
Time Frame: Baseline up to 7-10 days after the last dose of study drug (up to 32 days)
Population: Safety analysis set included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (800 mg): Severe Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 4 | 8 | 8 | 8 | 4
participants | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0

25. Secondary Outcome: Number of Participants With 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Criteria for abnormal ECG (12-lead) values were defined as: maximum PR interval >=300 millisecond (msec) and maximum increase of >=25 percent for baseline value of >200 msec and >=50% for baseline value of <=200 msec for PR interval, QRS interval >=200 msec; QT interval corrected using the Fridericia formula (QTcF) >=500 msec or increase of >45 msec.
Time Frame: Baseline up to 7-10 days after the last dose of study drug (up to 32 days)
Population: Safety analysis set included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (800 mg): Severe Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 4 | 8 | 8 | 8 | 4
participants | 0 | 3 | 0 | 0 | 3 | 1 | 4 | 4 | 2

26. Secondary Outcome: Number of Participants With Change From Baseline in Physical Examinations
Description: Physical examination included examination of the skin, eyes, ears, throat, neck, and cardiac, respiratory, gastrointestinal and musculoskeletal systems. The examination assessed the participants for any potential changes in physical status, as determined by the investigator. Any untoward findings identified on physical exams conducted after the administration of the first dose of study medication was captured as an adverse event.
Time Frame: Baseline, 7-10 days after the last dose of study drug
Population: Safety analysis set included all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (800 mg): Severe Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 1 | 4 | 8 | 8 | 8 | 4
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 7-10 days after the last dose of study drug (up to 32 days)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- PF-03709270 (1000 mg): Severe Renal: Participants with severe renal impairment received a single oral dose of PF-03709270 1000 mg tablet under fasted condition in second intervention period.
Arm/Group | CP-70,429 (800 mg): Normal Renal Function | CP-70,429 (800 mg): Mild Renal Impairment | CP-70,429 (800 mg): Moderate Renal Impairment | CP-70,429 (800 mg): Severe Renal Impairment | CP-70,429 (200 mg): Severe Renal Impairment | PF-03709270 (1000 mg): Normal Renal Function | PF-03709270 (1000 mg): Mild Renal Impairment | PF-03709270 (1000 mg): Moderate Renal Impairment | PF-03709270 (1000 mg): Severe Renal
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/1 | 1/4 | 0/8 | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 5/8 | 5/8 | 4/8 | 0/1 | 3/4 | 6/8 | 4/8 | 6/8 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-70,429 (800 mg): Normal Renal Function (N=8) | CP-70,429 (800 mg): Mild Renal Impairment (N=8) | CP-70,429 (800 mg): Moderate Renal Impairment (N=8) | CP-70,429 (800 mg): Severe Renal Impairment (N=1) | CP-70,429 (200 mg): Severe Renal Impairment (N=4) | PF-03709270 (1000 mg): Normal Renal Function (N=8) | PF-03709270 (1000 mg): Mild Renal Impairment (N=8) | PF-03709270 (1000 mg): Moderate Renal Impairment (N=8) | PF-03709270 (1000 mg): Severe Renal (N=4)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-70,429 (800 mg): Normal Renal Function (N=8) | CP-70,429 (800 mg): Mild Renal Impairment (N=8) | CP-70,429 (800 mg): Moderate Renal Impairment (N=8) | CP-70,429 (800 mg): Severe Renal Impairment (N=1) | CP-70,429 (200 mg): Severe Renal Impairment (N=4) | PF-03709270 (1000 mg): Normal Renal Function (N=8) | PF-03709270 (1000 mg): Mild Renal Impairment (N=8) | PF-03709270 (1000 mg): Moderate Renal Impairment (N=8) | PF-03709270 (1000 mg): Severe Renal (N=4)
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 4 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.